CLINICAL TRIAL: NCT00288522
Title: A Phase II, Single Centre, Randomized, Double-blind, Parallel and Placebo Controlled, Pilot Study to Evaluate the Efficacy and Safety of Somatuline Autogel 60mg in Patients With Active Thyroid-associated Ophthalmopathy of Moderate Intensity.
Brief Title: Lanreotide (Somatuline Autogel) in Thyroid-associated Ophthalmopathy Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-92-52030-164; 2004-003937-14 (EudraCT Number)
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Thyroid-Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — lanreotide

INTERVENTIONS:
Drug: Lanreotide (Autogel formulation). Duration of treatment - 3 injections, 1 every 28 days

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of 3 doses of Somatuline Autogel 60mg to control the muscle infiltration and edema, eyelid retraction and extraocular muscular contraction in patients with active thyroid-associated ophthalmopathy of moderate intensity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with autoimmune thyroid disease and whose centre's medical records confirm the presence of euthyroidism for at least two months before being included into the study
* Thyroid-associated ophthalmopathy diagnosed a minimum of six months before his/her participation in the study, well documented in the centre's medical records and based on the moderate intensity of thyroid-associated ophthalmopathy in the worst eye
* Patients whose ophthalmopathy activity has been demonstrated by a positive octreoscan

Exclusion Criteria:

* The patient presents compressive optical neuropathy signs which require immediate surgical treatment or suffers from serious intensity thyroid ophthalmopathy
* The patient has been treated with radio-iodine for his/her thyroid disturbance in the past 6 months
* The patient's thyroid-associated ophthalmopathy has been treated previously (except for drops and local measures) or is planned to be treated with radio-iodine or thyroidectomy for his/her autoimmune thyroid disease during the study or suffers from myopia, glaucoma or any other eye disease which could modify the ophthalmological progress
* The patient is a smoker of more than 5 cigarettes per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Extraocular muscle infiltration and edema exam by evaluating (at Day 0 and Weeks 4, 8 and 12): extraocular muscle size, proptosis and intraocular pressure (tonometry)
Eye inspection (at Day 0 and Weeks 4, 8 and 12): assessment of conjunctival injection presence, chemosis, cheratitis and eyelid edema; extrinsic muscle function evaluation and eyelid retraction

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Hospital General d'Alacant, Alicante, Spain